CLINICAL TRIAL: NCT04031638
Title: Prospective and Retrospective Thyroid Cancer Database
Brief Title: Thyroid Cancer Database
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: AB2015THYROID
Record Dates: First submitted 2019-07-01; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Patients With a Thyroid Tumor Who Received Radioactive Iodine Treatment
Keywords: Thyroid cancer, Iodine treatment
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radioactive Iodine treatment for thyroid cancer
  Interventions: Other: Radioactive Iodine treatment

INTERVENTIONS:
Other: Radioactive Iodine treatment — Patients with a thyroid tumor who received radioactive Iodine treatment.

SUMMARY:
Thyroid cancer database collects clinical and laboratory data from patients with a thyroid tumor who received radioactive Iodine treatment. This database only records information based on patients' medical files in a structured manner.

Thyroid database is used for retrospective non-interventional research projects.

ELIGIBILITY:
Inclusion Criteria:

* patients with a thyroid tumor (metastatic or not)
* patients who received radioactive Iodine treatment.
* age >= 18

Exclusion Criteria:

* Objection to collect medical data records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a thyroid tumor who received radioactive Iodine treatment in Centre Georges Francois Leclerc, Dijon, France
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient survival | 10 years
  Overall survival and evolution over years

SECONDARY OUTCOMES:
Collection of patient and treatment characteristics | 10 years
  Collection of patient and treatment characteristics over years, to set up prospective and retrospective studies

CONTACTS AND LOCATIONS:
Locations (1):
- Methodology, Biostatistics and Data Management, Dijon, France

IPD SHARING:
Plan to Share IPD: No